CLINICAL TRIAL: NCT01310556
Title: The Relationship Between Previously Unknown Glucose Metabolism Disorders and Coronary Artery Disease in Patients Suffering From Coronary Artery Disease
Brief Title: Unknown Glucose Metabolism Disorders In Patients With Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Gulhane School of Medicine, Dep. of Endocrinology and Metabolism
Other Study IDs: 12.05.2009-131-1068
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus
Keywords: OGTT; coronary artery disease
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- coronary artery disease: patients with coronary artery disease
  Interventions: Other: ogtt for patients with coronary artery disease

INTERVENTIONS:
Other: ogtt for patients with coronary artery disease — 75 g OGTT
  Other Names: no name

SUMMARY:
This study aimed to examine the prevalence of glucose metabolism disorders (GMD)in the patients with coronary artery disease and the relationship between different GMDs and coronary artery disease (CAD).

DETAILED DESCRIPTION:
Context: There are more than 220 million people diagnosed with diabetes mellitus (DM) in the world. DM is a serious risk factor for coronary artery disease (CAD). This study aimed to examine the prevalence of glucose metabolism disorders (GMD) in te patients with coronary artery disease and the relationship between different GMDs and CAD.

Settings: 230 patients with coronary artery disease and without any known GMDs were included the study. Coronary angiography was used to diagnose CAD. Patients were administered the 75 g Oral Glucose Tolerance Test (OGTT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease and who had no glucose metabolism disorders were included to study.

Exclusion Criteria:

* Patients who had previous GMDs, malignancies, chronic liver and kidney diseases, rheumatologic disorders, and a BMI higher than 35 kg/m2 were excluded from the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery disease and who had no glucose metabolism disorders.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Frequency of unknown glucose metabolism disorders in patients with coronary artery disease | 1 year
  Results: While GMDs were detected in 58.26% (n=134 patients) of CAD patients, 41.74% of them (n=96 patients) were found to have normal glucose metabolism.

SECONDARY OUTCOMES:
Fasting and 120 minute glucose levels have relation with vessels' stenosis. | 1 year
  Fasting glucose level was found to have a significant correlation with the total number of stenotic coronary vessels (p=0.0001) and the stenosis rate of all vessels . OGTT 120-minute glucose levels were found to have a significant correlation with the total number of stenotic coronary vessels and the stenosis rate of vessels with the exception of LAD.

CONTACTS AND LOCATIONS:
Overall Officials: Aydogan Aydogdu, MD, Study Director — Gulhane School of Medicine Ankara/Turkey
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)